CLINICAL TRIAL: NCT00544635
Title: The Effect Of Light On Scar Appearance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study personnel left institution before study completion.
Sponsor: Northwestern University (Other)
Responsible Party: Murad Alam, MD, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1253-010
Record Dates: First submitted 2007-10-12; First posted 2007-10-16 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Cutaneous Scars
MeSH Terms: interventions — Ultraviolet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): scars will be treated with light
  Interventions: Device: light
- B (Placebo Comparator): no intervention
  Interventions: Device: no intervention

INTERVENTIONS:
Device: no intervention — no intervention
  Arms: B
Device: light — scars will be treated with light
  Arms: A

SUMMARY:
The goal of this project is to examine the ability of light exposure to improve the appearance of cutaneous scars.

DETAILED DESCRIPTION:
Light would be efficacious in improving scar appearance due to its known effects on wound healing, acne, and its use for skin rejuvenation. Light interacts with cells and stimulates the production of new collagen and elastin. This same energy can be used to inhibit collagen formation and help improve scars.

ELIGIBILITY:
Inclusion Criteria:

* Have two lesions that have been selected for excision
* Have two cutaneous scars from previous excisions as part of a standard of care
* Subjects are in good health
* Subject has a willingness and the ability to understand and provide informed consent for the use of their tissue and communicate with the investigator

Exclusion Criteria:

* Pregnancy or lactation
* Subjects who are unable to understand the protocol or to give informed consent
* Subjects with mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-11; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Scar vascularity | 24 weeks
Scar pigmentation | 24 weeks
Scar thickness | 24 weeks
Scar length | 24 weeks
Scar width | 24 weeks
Scar surface area | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States